CLINICAL TRIAL: NCT04409093
Title: A Prospective, Randomized, Controlled Trial Evaluating the Utility of Eponychial Stents for Nail Re-growth in Nail Bed Injuries
Brief Title: Eponychial Stent Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-00355
Record Dates: First submitted 2020-05-21; First posted 2020-06-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Eponychial Stent; Nail Bed Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nail bed repair with eponychial sent (Experimental)
  Interventions: Procedure: Nail bed repair with eponychial sent
- Nail bed repair without eponychial stent (Active Comparator)
  Interventions: Procedure: Nail bed repair without eponychial stent

INTERVENTIONS:
Procedure: Nail bed repair with eponychial sent — The nail bed repair will be performed with 6-0 chromic suture material. After the nail bed repair, an eponychial stent will be secured under the eponychial fold with suture. The stent can be the native nail plate, suture container foil, or nonadherent gauze (i.e. Xeroform). If the injury avulsed the nail plate and the patient presents without it, either the foil from the suture wrapper/container or a piece of nonadherent gauze (i.e. Xeroform) will be used as a stent. A nonadherent sterile dressing will be applied to the digit, and each patient will be discharged with a 5-day course of cephalexin for prophylaxis against infection.
  Arms: Nail bed repair with eponychial sent
Procedure: Nail bed repair without eponychial stent — The nail bed repair will be performed with 6-0 chromic suture material. After the nail bed repair, an eponychial stent will not be secured under the eponychial fold. A nonadherent sterile dressing will be applied to the digit, and each patient will be discharged with a 5-day course of cephalexin for prophylaxis against infection.
  Arms: Nail bed repair without eponychial stent

SUMMARY:
The study design is a prospective, randomized, controlled trial evaluating the cosmetic and functional outcomes of nail bed repairs with and without eponychial stents. Patients presenting to a single institution with a finger tip injury requiring a nail bed repair will be initially evaluated in the emergency department. The purpose of the study will be explained to the patient, and informed consent for participation will be obtained. Patients will be randomly assigned to either the eponychial stent or no eponychial stent group based on the last digit of their assigned medical record number. Even-numbered patients will be randomized to the stent group and odd-numbered patients will be randomized to the no stent group. Demographic data will be obtained and recorded (age, gender, hand dominance, mechanism of injury, and past medical history). All patients will undergo a thorough clinical exam under digital nerve block followed by removal of the nail plate and thorough irrigation and debridement of devitalized tissue. The nail bed repair will be performed with 6-0 chromic suture material. After the nail bed repair, a stent (native nail, suture container foil, or nonadherent gauze) will or will not secured under the eponychial fold with suture depending on randomization. Laceration characteristic and time required to perform the procedure will be recorded. A nonadherent sterile dressing will be applied to the digit, and each patient will be discharged with a 5-day course of cephalexin for prophylaxis against infection. Follow-up evaluation will occur at 1 week, 1 month, 3 months, and 6 months. A each follow-up visit, patient-perceived functional outcome, cosmetic outcome, and level of pain will be assessed using a 10-point analog scale. Cosmetic results will also be evaluated by the examining physician using a validated physician-based outcome tool.

ELIGIBILITY:
Inclusion criteria:

1. Men and women, age > 18 years.
2. Patients with either nail plate avulsion and/or fracture with associated nail bed injury or subungal hematoma > 50% with intact nail plate.
3. Presentation within 8 hours of injury.
4. Being treated at NYU Langone Health or Jamaica Hospital Medical Center.
5. Willingness to participate in the study

Exclusion criteria:

1. Nail plate/bed injury secondary to bite wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Patient reported score on functional outcome scale (10-point analog scale) | after procedure: 1 week, 1 month, 3 months, and 6 months
  Mean score from all time points
  0 = complete loss of affected digit function during activities of daily living and recreational activities 10 = no functional limitation
Patient reported score on cosmetic outcome scale (10-point analog scale) | after procedure: 1 week, 1 month, 3 months, and 6 months
  Mean score from all time points
  0 = cosmetically unacceptable 10 = no perceived difference between treated finger and the same finger on the contralateral hand
Patient reported pain level on Visual Analog Scale (VAS) | after procedure: 1 week, 1 month, 3 months, and 6 months
  Mean score from all time points
  0 = no pain 10 = persistent finger pain during rest and activity
Physician reported cosmetic outcome | after procedure: 1 week, 1 month, 3 months, and 6 months
  Mean score from all time points
  Zook et al. Excellent = identical in appearance to the same finger on the contralateral hand Very good = 1 variation from identical, such as incomplete adherence, nail ridging, split nails, or eponychial deformity.
  Good = 2 minor variations from identical. Poor = more than 3 variations or 1 major variation from the same finger on the contralateral hand.

SECONDARY OUTCOMES:
Procedure time | 0-1 hour
  To determine the added time taken to perform the eponychial stent following nail bed repair

CONTACTS AND LOCATIONS:
Overall Officials: Nader Paksima, DO MPH, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - NYU Langone Orthopedic Hospital, New York, New York
  - Tisch Hospital, NYU Langone Health, New York, New York
  - Jamaica Hospital Medical Center, Richmond Hill, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [contact information for PI or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to ali.azad@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.